CLINICAL TRIAL: NCT05930509
Title: Home-based Non-invasive Brain Stimulation for Treatment-resistant Depression: Feasibility, Efficacy and Biomarker of Treatment Response
Brief Title: Home-based Non-invasive Brain Stimulation for Treatment-resistant Depression Feasibility, Efficacy and Biomarker of Treatment Response
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Guttmann (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Gabriele Cattaneo, Principal Investigator, Institut Guttmann
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Institut Guttmann
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Open clinical trial
Masking Description: All participants will receive the same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): tDCS stimulation
  Interventions: Device: Non-invasive transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Non-invasive transcranial direct current stimulation (tDCS) — Electrical stimulation

SUMMARY:
Depression has a yearly prevalence superior to 5%, but a 30% of patients cannot benefit of pharmacological treatment, resulting resistant to it.

Transcranial direct current stimulation, due to its reduced invasiveness and easy administration showed to be a useful technique to treat these cases, and it is now broadly used in clinical practice.

Moreover, thanks to technological advances, this treatment could be self-administered at home, reducing costs and improving scalability.

The aim of this study is to confirm the efficacy, safety and feasibility of a home-based intervention for treatment-resistant depression

To do this participants will perform a home-based tDCS intervention consisting of 30 minutes sessions, 5 days per week, for 4 weeks.

Results should provide critical knowledge regarding home-based therapies for the treatment of resistant depression and evidence on brain mechanisms underlying response to non-invasive brain stimulation.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a highly disabling pathology with an important prevalence along the whole lifespan. Its global prevalence is around 5% of the population and it has been estimated that depression represents the third cause of worldwide disability causing an enormous social and economic impact.

While a significant proportion of patients with MDD show clinical responses to first line pharmacological interventions, almost 30% of cases exhibit resistance to medications, and fail to gain remission of symptoms when administered with antidepressants.

This condition, termed treatment-resistant depression (TRD), defines patients where treatment with two or more products of different pharmacological classes used for a sufficient length of time at an adequate dose, fails to induce a clinically meaningful effect (inadequate response).

TRD worsens the personal, social, and economic impact of depression and TRD patients, compared to non-TRD patients, reported reduced quality of life, reduced physical and mental health, presenting important impairments in daily life activities. Furthermore, for these patients, healthcare resources and costs are also significantly higher.

To treat these patients in the last decades various alternative therapeutic approaches have been developed. Between them non-invasive brain stimulation (NIBS) demonstrated to be a safe and effective procedure that successfully reduces and mitigates major depression symptoms.

Amongst the different techniques, transcranial direct current stimulation (tDCS) is one of the more studied and promising approaches, as it can modulate cortical activity related to cognitive control dysfunction in MDD.

In tDCS, surface electrodes (anode and cathode) inject low-amplitude direct current through the scalp to modulate brain activity and excitability, with regulatory effects impacting not only the brain areas stimulated but also at the level of brain networks, and therefore with the potentiality of 'optimizing' the balance between integration and segregation of associated functions, commonly observed in neuropsychiatric conditions.

In recent years, tDCS showed to be safe and generally well-tolerated when appropriate safety guidelines are followed, and has demonstrated a moderate but consistent effect in depression treatment.

Crucially, recent tDCS systems are highly portable and easy to set-up, with the possibility to be configurated remotely, potentially allowing the administration of remotely supervised non-pharmacological treatments at home, facilitating long duration treatments adherence.

Recently, scientific interest in the application of home-based tDCS to a variety of clinical conditions has increased progressively, and regarding to depression.

This potentially represents a very relevant step forward in the treatment of TRD, making it very scalable and highly feasible for people living far from clinical facilities, with displacement difficulties or considering exceptional situations as the COVID-19 pandemic that on one hand absorbed most healthcare resources and on the other impose to people to eliminate or reduce mobility.

Aim:

The aim of this study is to confirm the efficacy and feasibility of a home-based intervention for treatment-resistant depression

Hypothesis:

The specific hypothesis is that it is feasible and effective to implement a self-administered home-based therapeutic intervention to reduce or eliminate depressive symptoms.

Material and Methods:

Design

The investigators will implement an home-based brain stimulation treatment using tDCS in people suffering from TRD. The stimulation will be administered in collaboration with a familiar (companion) that will participate, together with the patients, in a training on tDCS administration before the beginning of the treatment. Moreover, the treatment will be preceded and followed by pre and post assessments.

Participants

The investigators will enroll 40 participants, over 18 years old. Sample size has been calculated considering the effect size of the few previous studies investigating the modulatory effect of non-invasive brain stimulation on behavioral outcomes of depression (Hedge's g = 0.3-0.76).

Sample sizes needed for the type of analysis presented in the "statistical approach section" (F statistics as repeated measure ANOVA, logistic and linear regressions, etc..), considering alpha=0.05 and statistical power (1-beta) =0.80, for the interventional study to be conducted is estimated to be of 40 participants, considering a 10-15% drop-out.

Companion training

Before beginning the intervention the investigators will undertake a first in-person training session, followed by remote training and supervision program, for companions that will administer the stimulation. These training sessions will have the aim to instruct about ,and assure, the correct administration of the stimulation.

The program will be based on three main pillars: an in-depth training curriculum about tDCS and instructions on how to administer the stimulation, a set of remote practice sessions hosted by trained research staff for study companions to promptly apply the knowledge and skills derived from the training curriculum, and an on-demand remote assistance infrastructure to provide additional support and guidance to study companions as needed.

Pre-Post assessment

Before and after the stimulation protocol participants will be administered with questionnaires and scales to evaluate our main outcomes.

Efficacy outcomes

Participants will be administered with the Montgomery-Åsberg Depression Rating Scale (MADRS), the Beck Depression Inventory, the Hamilton Depression Rating Scale and the patient participant-rated Quick Inventory of Depressive Symptomatology. Moreover, participants will also be cognitively assessed with a cognitive screening and regarding their quality of life with the administration of the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form. The investigators also administer a cognitive screening using the "Guttmann Cognitest"digital solution, and the Montreal Cognitive Assessment (MOCA) for self-administered cognitive testing.

Feasibility outcomes

To assess feasibility of the treatment the investigators will evaluate the adherence to the intervention in terms of compliance of scheduled sessions measuring the decreasing of electrode impedance and the number of aborted sessions due to high electrodes impedance.

tDCS study protocol: general montage and configuration procedures

Stimulation will consist of 20 sessions over three consecutive weeks (from Monday to Friday), each session lasting for 30 minutes, following a protocol broadly used in various clinical centers and approved for depression treatment.

The stimulation will target the left dorsal lateral prefrontal cortex (L-DLPFC), consistently previously identified as target for tDCS depression treatment.

Current will be supplied in a constantly for 30 minutes and will be initially increased and finally decreased in a 30 s ramp-up and ramp-down fashion. All stimulation parameters adhere to general transcranial electrical stimulation current safety criteria guidelines and for safety issues, the maximum current delivered will be 2 ma.

Stimulation will be delivered via "Sooma tDCS™" medical device, used by healthcare professionals worldwide. It has acquired e.g. CE, Health Canada, MDA, HSA, TGA and COFEPRIS approvals for the treatment of depression. "Sooma tDCS™" devices are manufactured in Finland under ISO 13485. This device has been designed to be very easy to use anywhere having a single control button that is used to start and pause the stimulation. Everything else is automated and consequently, the presence of a medical professional is not required during the treatment sessions and patients may perform the therapy from the comfort of their home. In addition, with the help of a cloud-based software suit the physician could follow app treatment progress instantly .

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria and be diagnosed by a Psychiatrist for MDD, according to the Diagnostic and Statistical Manual of Mental Disorders
* Score at least 20 on the Montgomery-Åsberg Depression Rating Scale
* Be stable enough to participate in the study without risk for safety.
* Live with an adult with computer skills and willingness to learn how to use tDCS.

Exclusion criteria:

* Present other psychiatric conditions or neurological disorders
* Abuse of alcohol or drugs
* Pregnancy
* Present any contraindication for tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | immediately after the intervention
  Number of session completed
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | immediately after the intervention
  Incidences related with the stimulation

SECONDARY OUTCOMES:
Changes in the Montgomery-Åsberg Depression Rating Scale | baseline and immediately after the intervention
  depression scale scoring from 0 to 60, where higher scores represent more severe depression
Changes in the Beck Depression Inventory | baseline and immediately after the intervention
  depression scale scoring from 0 to 63, where higher scores represent more severe depression
Changes in the Hamilton Depression Rating Scale | baseline and immediately after the intervention
  depression scale scoring from 0 to 68, where higher scores represent more severe depression
Changes in the Quick Inventory of Depressive Symptomatology | baseline and immediately after the intervention
  depression scale scoring from 0 to 27, where higher scores represent more severe depression
Changes in the Montreal Cognitive Assessment | baseline and immediately after the intervention
  cognitive scale scoring from 0 to 30 where higher scores represent better cognitive functioning
Changes in the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form | baseline and immediately after the intervention
  QoL scale scoring from 0 to 30, where higher scores represent better cognitive functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Guttmann Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided